CLINICAL TRIAL: NCT02956304
Title: " Effect of Affordance of Objects on the Memory: Study in Transcranial Magnetic Stimulation " (SIMULANG-TMS)
Brief Title: " Effect of Affordance of Objects on the Memory: Study in Transcranial Magnetic Stimulation "
Acronym: SIMULANG-TMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: University of Paris 5 - Rene Descartes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: D15-P13
Record Dates: First submitted 2016-07-20; First posted 2016-11-07 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Healthy
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group iTBS-cTBS-SHAM (Other): PMv stimulation (iTBS) at session 2, PMv inhibition (cTBS) at session 3, and control (SHAM) at session 4
  Interventions: Other: PMv stimulation (iTBS); Other: PMv inhibition (cTBS); Other: Control (SHAM)
- Group iTBS-SHAM-cTBS (Other): PMv stimulation (iTBS) at session 2, control (SHAM) at session 3, and PMv inhibition (cTBS) at session 4
  Interventions: Other: PMv stimulation (iTBS); Other: PMv inhibition (cTBS); Other: Control (SHAM)
- Group cTBS-iTBS-SHAM (Other): PMv inhibition (cTBS) at session 2, PMv stimulation (iTBS) at session 3, and control (SHAM) at session 4
  Interventions: Other: PMv stimulation (iTBS); Other: PMv inhibition (cTBS); Other: Control (SHAM)
- Group cTBS-SHAM-iTBS (Other): PMv inhibition (cTBS) at session 2, control (SHAM) at session 3, and PMv stimulation (iTBS) at session 4
  Interventions: Other: PMv stimulation (iTBS); Other: PMv inhibition (cTBS); Other: Control (SHAM)
- Group SHAM-iTBS-cTBS (Other): control (SHAM) at session 2, PMv stimulation (iTBS) at session 3, and PMv inhibition (cTBS) at session 4
  Interventions: Other: PMv stimulation (iTBS); Other: PMv inhibition (cTBS); Other: Control (SHAM)
- Group SHAM-cTBS-iTBS (Other): control (SHAM) at session 2, PMv inhibition (cTBS) at session 3, and PMv stimulation (iTBS) at session 4
  Interventions: Other: PMv stimulation (iTBS); Other: PMv inhibition (cTBS); Other: Control (SHAM)

INTERVENTIONS:
Other: PMv stimulation (iTBS) — PMv stimulation (iTBS)
Other: PMv inhibition (cTBS) — PMv inhibition (cTBS)
Other: Control (SHAM) — Control (SHAM)

SUMMARY:
The purpose of this study is determine the involvement of motor system in the memory of manipulable objects. The idea is to stimulate the ventral premotor cortex with transcranial magnetic stimulation to see whether this stimulation will affect memory of manipulable objects.

DETAILED DESCRIPTION:
Embodied cognition claims that representations shares processing resources with sensorimotor systems. More specifically, it has been proposed that language comprehension relies on internal simulation of the meaning. For instance, numerous studies have shown that the processing of action-related concepts involve a motor activation similar to when the action is actually performed. However, even if those studies show clearly that action-related concepts involve a motor activation, such activations may be incidental to the activation of their representations, rather than part of it. Another way to show that this motor component takes part in the representation of manipulable objetcs is to investigate whether an impairment of motor system would impair the memory of manipulable object. In this study, investigators will use Transcranial Magnetic Stimulation (TMS) to stimulate ventral premotor cortex (PMv) to see whether this stimulation will affect memory of manipulable objects, but not memory of nonmanipulable objects. For this purpose, three TMS conditions will be assessed: cTBS to inhibit the motor cortex, iTBS to excite the motor cortex, and a SHAM condition as control.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 35 years
* Right-handers (score between 70 and 100 on the scale of Edinburgh)
* Native language : French
* Not depressed (score lower than 14 in the BDI)
* health insurance
* Consent

Exclusion Criteria:

* Psychiatric family history up to the second degree
* Medical treatment, in particular psychotropic being able to affect the memory and the attention
* view or hearing disorders (not compensated)
* neurological histories (epilepsy, alcoholism in particular) or psychiatric or important memory complaints
* Contraindications for the SMT
* contraindications in the MRI

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Number of objects affordants and of objects not - affordants reminded | 1 week
  Measure of the number of objects affordants and of objects not - affordants reminded according to if the stimulation is in PMv or control
Number of objects affordants and of objects not - affordants reminded | 2 weeks
  Measure of the number of objects affordants and of objects not - affordants reminded according to if the stimulation is in PMv or control
Number of objects affordants and of objects not - affordants reminded | 3 weeks
  Measure of the number of objects affordants and of objects not - affordants reminded according to if the stimulation is in PMv or control

SECONDARY OUTCOMES:
Number of object reminded | 1 week
  Measure of the number of objects affordants and of objects not - affordants reminded according to if the stimulation is excitation or control
Number of object reminded | 2 weeks
  Measure of the number of objects affordants and of objects not - affordants reminded according to if the stimulation is excitation or control
Number of object reminded | 3 weeks
  Measure of the number of objects affordants and of objects not - affordants reminded according to if the stimulation is excitation or control

CONTACTS AND LOCATIONS:
Overall Officials: Pascale PIOLINO, Study Director — University of Paris 5 - Rene Descartes; Benoit CREPON, MD, Study Director — CHSA
Locations (1):
- Centre de Recherche Clinique (CRC) - CHSA, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided